CLINICAL TRIAL: NCT00057395
Title: A Phase I/II Study of Aroplatin™ in Patients With Advanced Solid Malignancies
Brief Title: A Safety and Effectiveness Study of Aroplatin in Patients With Advanced Solid Malignancies
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aronex Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-726-04
Record Dates: First submitted 2003-04-01; First posted 2003-04-02 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-04

CONDITIONS: Esophageal Neoplasms; Hepatocellular Carcinoma; Colorectal Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Neoplasms
Keywords: Esophageal Neoplasms; Esophagus Neoplasm; Esophagus Cancer; Esophageal Cancer; Esophageal Tumors; Esophagus Tumors; Neoplasms, Esophageal; Hepatocellular Carcinoma; Carcinoma, Hepatocellular; Hepatoma; Colorectal Neoplasms; Colorectal Cancer; Colorectal Carcinoma; Colorectal Tumor; Neoplasms, Colorectal; Ovarian Neoplasms; Ovary Neoplasms; Ovary Cancer; Ovary Carcinoma; Ovarian Cancer; Ovarian Carcinoma; Neoplasms, Ovarian; Pancreatic Neoplasms; Pancreatic Cancer; Pancreas Neoplasms; Pancreas Cancer; Neoplasms, Pancreatic; Neoplasms, Pancreas; and other solid tumors
MeSH Terms: conditions — Esophageal Neoplasms; Carcinoma, Hepatocellular; Colorectal Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Neoplasms | interventions — bis-neodecanoato-1,2-diaminocyclohexaneplatinum(II)

INTERVENTIONS:
Drug: Aroplatin (Liposomal NDDP, L-NDDP)

SUMMARY:
To determine the rate of response and the duration of the response following therapy with Aroplatinin patients with advanced solid malignancies.

DETAILED DESCRIPTION:
Primary Objective:

* Determine response rate (RR; complete and partial response [CR, PR]) and duration after therapy with Aroplatin™ in patients with advanced solid malignancies.

Secondary Objective:

* Determine the safety and tolerability of Aroplatin

ELIGIBILITY:
Inclusion Criteria:

* Advanced solid malignancies;
* Amenable to therapy with DACH platinum agents;
* Measurable disease (RECIST criteria);
* ECOG performance score of 0-2;
* Adequate hematopoietic, liver and renal function;
* Adequate cardiac function (maximum of class II, NYHA);
* Women of childbearing potential must have a negative urine or serum pregnancy test;
* Signed written informed consent;
* Subjects must be willing to be followed during the course of treatment/observation and follow-up.

Exclusion Criteria:

* No other active malignancies;
* No prior therapy with oxaliplatin;
* No known brain metastases;
* Active, uncontrolled infection or other serious medical illnesses;
* Not using or have used any investigational therapy during four weeks before start of protocol treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40

CONTACTS AND LOCATIONS:
Locations (1):
- John Wayne Cancer Institute, Santa Monica, California, United States